CLINICAL TRIAL: NCT07309354
Title: The Effects of Tizanidine on Acoustic Reflex
Brief Title: Tizanidine and Acoustic Reflex
Acronym: TIZ-AR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TIZAR470; USAKBAP2025671 (Other Grant/Funding Number: Usak University)
Record Dates: First submitted 2025-12-15; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Reflex, Acoustic; Hearing
Keywords: tizanidine; acıustic reflex; hearing
MeSH Terms: interventions — tizanidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tizanidine Pre-Post Evaluation (Experimental): Participants in this single-arm study will receive tizanidine 6 mg orally once daily for 1 week. Standardized audiological testing, including tympanometry and acoustic reflex measurements, will be performed twice: once before starting tizanidine and again at the end of the treatment period. Pre- and post-treatment acoustic reflex thresholds and response patterns will be compared within the same participants.
  Interventions: Drug: Tizanidine

INTERVENTIONS:
Drug: Tizanidine — Participants will receive tizanidine 6 mg orally once daily for 1 week. Standardized audiological testing, including tympanometry and multifrequency acoustic reflex measurements, will be performed before starting treatment and on day 7 at the end of the treatment period to evaluate changes in acoustic reflex thresholds and response patterns.

SUMMARY:
The goal of this clinical trial is to learn how the muscle relaxant tizanidine affects the acoustic reflex in adults. The acoustic reflex is a natural protection system of the ear that helps reduce the impact of loud sounds. It is not known whether tizanidine changes how this reflex works.

The main question this study aims to answer is:

Does taking tizanidine for 1 week change acoustic reflex thresholds in the same person, when comparing before and after treatment? Participants who receive tizanidine will undergo hearing and acoustic reflex tests before treatment and again at the end of the treatment period.

DETAILED DESCRIPTION:
Tizanidine is a commonly used muscle relaxant prescribed for musculoskeletal pain. Its relaxing effect on body muscles is well known. However, it is not clear whether tizanidine also affects the small muscle in the middle ear that is responsible for the acoustic reflex.

The acoustic reflex is a natural protection system of the ear. When a loud sound occurs, a tiny muscle called the stapedius contracts. This contraction reduces the amount of sound energy that reaches the inner ear and helps protect the inner ear and hearing nerve from acoustic damage. If this reflex does not work properly, a person may become more sensitive to loud sounds and may be more vulnerable to noise-related ear injury.

Only a few studies have looked at how muscle relaxant medicines influence the acoustic reflex, and most of them focused on drugs used during anesthesia. There is very little information about tizanidine, which is used in daily clinical practice for muscle and joint pain. Because of this gap, it is important to understand whether tizanidine changes the strength or timing of the acoustic reflex.

This single-arm clinical study will follow adults who are already planned to receive tizanidine as part of their treatment. Participants will take tizanidine 6 mg by mouth once a day for 1 week. Hearing and acoustic reflex tests will be done twice: once before starting tizanidine and again at the end of the treatment period. The same standardized audiological methods will be used at both time points, including tympanometry and acoustic reflex measurements in both ears.

The main goal is to compare the acoustic reflex measurements before and after tizanidine treatment in the same participants. By looking at changes in acoustic reflex thresholds, amplitudes, and response patterns, the study aims to show whether tizanidine has a measurable effect on stapedius muscle function. If the results suggest that tizanidine weakens or delays the acoustic reflex, this could mean that patients taking tizanidine may need to be more careful about exposure to loud noise during treatment. The findings may help clinicians better understand the auditory safety of muscle relaxant therapy and guide practical advice for patients.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation and ability to provide informed consent
* Age 18 years or older
* Currently receiving tizanidine 6 mg once daily as part of clinical care
* No active middle ear disease that could affect tympanometric or acoustic reflex measurements
* No chronic neuromuscular disease
* Ability to complete audiological testing

Exclusion Criteria:

* Refusal to participate
* Withdrawal of consent at any time
* Age under 18 years
* Presence of any ear condition that affects the acoustic reflex (e.g., otitis media, tympanic membrane perforation, otosclerosis)
* Presence of chronic neuromuscular disease
* Current alcohol or substance use disorder
* Any condition preventing completion of acoustic reflex or tympanometry testing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Change in Acoustic Reflex Threshold | Baseline (before treatment) and Day 7 (end of treatment)

CONTACTS AND LOCATIONS:
Locations (1):
- Uşak University Faculty of Medicine, Uşak, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to institutional restrictions on the external sharing of personal health information.